CLINICAL TRIAL: NCT04964050
Title: An Open-label, Randomized Three Period, Three Sequence, Partially Replicated Crossover Bioequivalence Study of Two Oral Formulations of Captopril/Hydrochlorothiazide 50/25 mg Tablets in Healthy Adult Participants Under Fasting Conditions
Brief Title: A Bioequivalence Study Between Capozide Versus ACE-Hemmer-ratiopharm in Healthy Adult Participants Under Fasting Conditions
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Internal sponsor decision to terminate project prematurely based on a waiver granted by Egypt EDA (Egyptian drug authority). No subjects were enrolled.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 213049
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteers
Keywords: ACE-Hemmer-Ratiopharm; Bioequivalence; Capozide; Captopril/Hydrochlorothiazide
MeSH Terms: interventions — captopril, hydrochlorothiazide drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment sequence TRR (Experimental): Participants will receive Capozide (T) in period 1 followed by ACE-Hemmer-Ratiopharm (R) in period 2 followed by ACE-Hemmer-Ratiopharm (R) in period 3.
  Interventions: Drug: Capozide; Drug: ACE-Hemmer-Ratiopharm
- Treatment sequence RTR (Experimental): Participants will receive ACE-Hemmer-Ratiopharm (R) in period 1 followed by Capozide (T) in period 2 followed by ACE-Hemmer-Ratiopharm (R) in period 3.
  Interventions: Drug: Capozide; Drug: ACE-Hemmer-Ratiopharm
- Treatment sequence RRT (Experimental): Participants will receive ACE-Hemmer-Ratiopharm (R) in period 1 followed by ACE-Hemmer-Ratiopharm (R) in period 2 followed Capozide (T) by in period 3.
  Interventions: Drug: Capozide; Drug: ACE-Hemmer-Ratiopharm

INTERVENTIONS:
Drug: Capozide — Capozide will be administered as per the treatment sequence.
Drug: ACE-Hemmer-Ratiopharm — ACE-Hemmer-Ratiopharm will be administered as per the treatment sequence.

SUMMARY:
This is a bioequivalence study to compare Capozide (test product [T]) to ACE-Hemmer-ratiopharm (reference product[R]) produced by Ratiopharm GmbH Germany in healthy adult participants under fasting conditions.

ACE-Hemmer-ratiopharm®is the registered trademark of Ratiopharm GmbH Germany.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 50 years of age inclusive, at the time of signing the informed consent.
* Participant does not have a known allergy to the drug under investigation, any of its ingredients or any other related drugs.
* Normal vital signs after up to 10 minutes resting in supine position or 2 minutes in sitting position: 100 millimeters of mercury (mmHg) less than or equal to (<=) systolic blood pressure (SBP) <130 mmHg; 70 mmHg <= diastolic blood pressure (DBP) <90 mmHg; 60 beats per minute (bpm) <=Pulse rate (HR) <=100 bpm.
* Normal standard 12-lead ECG after 10 minutes resting in supine position in the following ranges; 120 microseconds (ms)<PR<220 ms, QRS<120 ms, QTc<=450 ms, and normal ECG tracing unless the Investigator considers an ECG tracing abnormality to be not clinically relevant.
* Laboratory parameters within the normal range (or defined screening threshold for the Investigator site), unless the Investigator considers an abnormality to be clinically irrelevant for healthy participants; however serum creatinine, alkaline phosphatase, hepatic enzymes (aspartate aminotransferase, alanine aminotransferase) should not exceed 1.25 times the upper laboratory normal, and total bilirubin should not exceed the upper laboratory normal. Laboratory tests are performed not longer than two weeks before the initiation of the clinical study).
* Body weight on 45 kilograms (kg) or more and body mass index (BMI) within the range 18.5 -30 kg per meter square (kg/m^2) (inclusive).
* Healthy Adult, male and female (woman of non-childbearing potential [WONCBP])
* Male participants are eligible to participate if they agree to the following during the study intervention period and for at least 30 days after the last dose of the study drug. Refrain from donating sperm PLUS, either be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR Must agree to use contraception/barrier as detailed below: Agree to use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential who is not currently pregnant, agree to use a male condom when engaging in any activity that allows for passage of ejaculate to another person. Contraceptive use by Men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. b) Female Participant is eligible to participate if she is a WONCBP. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy. Female participants must use a double contraception method including a highly effective method of birth control, except if she has undergone sterilization at least 3 months earlier or is postmenopausal.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular or infectious disease, or signs of acute illness, lactose intolerance.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* Blood donation, any volume, within 3 months.
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in SBP greater than or equal to (>=)30 mmHg within 3 minutes when changing from supine to standing position.
* Presence or history of drug hypersensitivity, participants with known hypersensitivity to any component of the investigational medicinal product (IMP) formulation or allergic disease diagnosed and treated by a physician. Participants who have previously demonstrated hypersensitivity to hydrochlorothiazide or to any sulfonamide-derived drugs.
* History of drug or alcohol abuse. History of regular alcohol consumption within one year of the study defined as: an average weekly intake of >14 drinks. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 milliliters [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Smoking regularly more than 5 cigarettes or equivalent per week, unable to stop smoking during the study (occasional smoker can be enrolled). Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses [average 100 mL] per day).
* Use of any prescribed medication, over the counter (OTC) medicines or medicinal products during the last two weeks preceding the first dosing and until discharge from the study.
* Participation in a bioequivalence study or in a clinical study within the last 60 days before first study drug administration.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis B core antibodies (anti-HBc Ab) if compound having possible immune activities, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab).
* Positive result on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
* Participants with a history of allergy or bronchial asthma or systemic lupus erythematosus.
* Participant who has results of laboratory tests which are outside the normal range or hemoglobin (Hb) or red blood cell (RBC) indices (mean corpuscular volume [MCV], mean corpuscular hemoglobin [MCH] and mean corpuscular hemoglobin concentration [MCHC]) with deviation outside 5% of the reference range. (Laboratory tests are performed not longer than two weeks before the initiation of the clinical study).
* Participants who have been on a specific/special diet during the 4 weeks before screening and who cannot agree to eat the set clinical food menu during the study.
* Participants that have a current active Coronavirus disease 2019 (COVID-19) infection, either laboratory confirmed or according to the investigator's medical judgement.
* Participants known to be in contact with active COVID-19 positive individuals within the past 14 days.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-21 (Estimated); Primary Completion 2022-05-26 (Estimated); Study Completion 2022-05-26 (Estimated)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of Captopril and Hydrochlorothiazide (HCTZ) | Up to 3 weeks
Area under the concentration-time curve from administration extrapolated to the last time of quantifiable concentration (AUC[0-t]) of Captopril and HCTZ | Up to 3 weeks
Area under the concentration-time curve from time zero extrapolated to infinite time (AUC[0-inf]) of Captopril and HCTZ | Up to 3 weeks

SECONDARY OUTCOMES:
Time to reach Cmax (Tmax) of Captopril and HCTZ | Up to 3 weeks
Terminal elimination halftime (t1/2) of Captopril and HCTZ | Up to 3 weeks
Terminal elimination rate constant (lambda-z) of Captopril and HCTZ | Up to 3 weeks
Percentage of AUC(0-inf) obtained by extrapolation (%AUCex) of Captopril and HCTZ | Up to 3 weeks
Number of participants with adverse events (AE) serious AEs | Up to 3 weeks
Number of participants with abnormal hematology and biochemistry parameters | Up to 3 weeks
Number of participants with abnormal electrocardiograms (ECGs) and vital signs findings | Up to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com